CLINICAL TRIAL: NCT04308707
Title: Breaking Bad News Skills of Doctors and Residents in Anesthesia and Surgical Specialties in Spain: a Cross-sectional Survey
Brief Title: Breaking Bad News Skills of Doctors and Residents in the Surgical Setting
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Enrique Carrero, MD, PhD, Senior Consultant in and Professor Anesthesiology, Hospital Clinic of Barcelona
Other Study IDs: BBNS-SS
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Communication Research; Patient Satisfaction; Communication Programs; Doctor Patient Relation
Keywords: Breaking bad news; Communication skills; Surveys and Questionnaires; Health Knowledge, Attitudes, Practice; Anesthesiology; Specialties, Surgical
MeSH Terms: conditions — Patient Satisfaction; Communication; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical specialties
  Interventions: Other: Breaking bad news skills
- Anesthesiology
  Interventions: Other: Breaking bad news skills

INTERVENTIONS:
Other: Breaking bad news skills — Communication skills analyzed by a specialized questionnaire designed from a Breaking bad news protocol developed in 2018-2019 in Barcelona.

SUMMARY:
Breaking bad news is a very stressful and difficult situation for health care professionals, especially clinical doctors and surgeons. Acquiring skills for this sort of communication is very important due to the large volume of times that these professionals will have to deal with it and because it can affect the doctor-patient relationship forever.

The objective of this study is to evaluate the skill of surgeons and residents in surgical specialties in breaking bad news to patients and families across Spanish hospitals. This will be done by analyzing the subjects in terms of their knowledge and experience using a specialized questionnaire based on breaking bad news protocol, designed in the "Hospital Sant Joan de Déu" Children's hospital in Barcelona.

ELIGIBILITY:
Inclusion Criteria:

- Doctors working in the Surgical Setting that accept and answer the specialized questionnaire.

Exclusion Criteria:

* Questionnaire answered out of the time-frame
* Incomplete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents and Doctors specialized in surgical specialties or anesthesiology.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of times having to communicate a bad new in the last year. | Two months
  Question on our questionnaire. The answer will be a number, expected to be from 0 to 200, approximately.
Number of hours in training in communication and breaking bad news skills. | Two months
  Question on our questionnaire. The answer will be the number of hours of professional training in the specific field of communication to patients.
Self-evaluation of the skills in breaking bad news and their self-perceived quality. | Two months
  In the self-administered questionnaire, 21 questions reflect specific and important items in communication designed from "La Primera notícia", a Breaking bad news protocol designed I the pediatric hospital "Hospital Sant Joan de Déu" in Barcelona.
  Data will be analyzed using GraphPad.
Knowledge of Second victim concept | Two months
  Direct question in our questionnaire: we ask the health-care professionals to define the Second victim concept.

SECONDARY OUTCOMES:
Where have the professionals acquired their skills in breaking bad news if they have not taken a training program? | Two months
  Question on our questionnaire. Possible answers are:
  * With the observation of peers and seniors.
  * Studying by themselves from books and papers.
  * Studying by themselves from videos and other internet content.
  * With the experience of years of working.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic of Barcelona, Hospital Uiversitari Mútua de Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided